CLINICAL TRIAL: NCT04901338
Title: Cytokine Hemoadsorption in ECMO Patients
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Jernej Berden, Jernej Berden, MD, PhD, University Medical Centre Ljubljana
Other Study IDs: Haemoadsorption ECMO
Record Dates: First submitted 2021-05-12; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: SIRS; Cytokine Storm; Cardiogenic Shock; Cardiac Arrest; Septic Shock; ARDS, Human
Keywords: Hemoadsorption; ECMO; SIRS; ARDS; Post-resuscitation syndrome; ECPR
MeSH Terms: conditions — Cytokine Release Syndrome; Shock, Cardiogenic; Heart Arrest; Shock, Septic; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Veno-arterial ECMO patients: Patients with severe SIRS post extracorporeal cardiopulmonary resuscitation (ECPR) or accompanying cardiogenic shock who were treated with hemoadsorption.
- Veno-venous ECMO patients: Patients with refractory septic shock on VV ECMO who were treated with hemoadsorption.

SUMMARY:
Cytokine hemoadsorption is a novel therapy used to improve outcome in critically ill patients with a dysregulated cytokine response and hemodynamic instability. Patients on extracorporeal membraneous oxygenation (ECMO) often develop severe systemic inflammatory response syndrome (SIRS). Cytokine removal using different types of hemoadsorption devices is believed to block the vicious circle of inflammation dysregulation when other basic therapeutic measures fail. To date there are very limited reports on ECMO and cytokine hemoadsorption combination therapy. The aim of this retrospective study is to evaluate feasibility and effectiveness of hemoadsorption in veno-arterial and veno-venous ECMO patients.

ELIGIBILITY:
Inclusion Criteria:

* VA/VV ECMO
* hemoadsorption
* Age ≥ 18 years

Exclusion Criteria:

* no additional exclusion criteria after being eligible for ECMO

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on VA ECMO or VV ECMO treated with hemoadsorption
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Haemodynamic stabilization | Within 12 hours after hemoadsorption
  Decreased need for vasopressors according to vasoactive-inotropic score and increase in mean arterial pressure

SECONDARY OUTCOMES:
Lactate, interleukin-6, C-reactive protein and procalcitonin clearance | Within 12 hours after hemoadsorption
Weaning from ECMO | from day of ECMO-implant for every 24 hours until date of weaning or death, whichever came first, assessed up to 90 days
ICU length of stay | from day of ICU-admission for every 24 hours until date of discharge or death, whichever came first, assessed up to 90 days
Hospital mortality | from day of hospital admission until date of discharge or death, whichever came first, assessed up to 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Ljubljana, Ljubljana, Slovenia